CLINICAL TRIAL: NCT06990750
Title: Insufflation Pressure and Postoperative Pain After Single Port Robotic Sacrocolpopexy
Brief Title: Single Port Insufflation RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB23-1711
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain Score
Keywords: insufflation pressure; postoperative pain; surgeon visualization; robotic sacrocolpopexy; single port sacrocolpopexy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pressure (Active Comparator): Insufflation pressure set to 15 mmHg (standard pressure).
  Interventions: Procedure: 15 mmHg
- Experimental Pressure (Experimental): Insufflation pressure set to 12 mm Hg (experimental pressure)
  Interventions: Procedure: 12 mmHg

INTERVENTIONS:
Procedure: 15 mmHg — Insufflation pressure was set to 15 mm Hg at the time of single port robotic sacrocolpopexy.
  Other Names: Standard insufflation pressure
  Arms: Standard pressure
Procedure: 12 mmHg — Insufflation pressure was set to 12 mm Hg at the time of single port robotic sacrocolpopexy.
  Other Names: Experimental insufflation pressure
  Arms: Experimental Pressure

SUMMARY:
The goal of this clinical trial is to learn if decreasing insufflation pressure during minimally invasive single port robotic sacrocolpopexy improved postoperative pain without impacting surgeon intraoperative visualization. The main question it aims to answer is:

Does minimally decreasing insufflation pressure improve postoperative pain?

Researchers will compare standard insufflation pressure (15 mmHg) to experimental insufflation pressure (12 mmHg) to see if it insufflation pressure impacts patient's postoperative pain.

Once a participants agrees to participate in our study, they will receive either standard or experimental pressure at the time of surgery. Postoperative pain scores in the postoperative anesthesia care unit and at postoperative day 1 and 14 visits will be recorded. Participants will also be asked to complete the Patient Global Impression of Improvement at the 14 day visit.

DETAILED DESCRIPTION:
This was a double-blinded, randomized control trial of women undergoing single port robotic sacrocolpopexy with intraperitoneal insufflation pressure set to 15 mm Hg (standard pressure) or 12 mm Hg (experimental pressure). Participants were randomized in a 1:1 ratio. Randomization was performed by an unblinded research coordinator with stratification by concomitant hysterectomy. Robotic surgeries were performed with the DaVinci single port robotic system, which supports the use of an 8-mm AirSeal port. Preoperative pain score (2 hours prior to surgery) were documented by a member of the research team. The operating room circulating nurse set the insufflation pressure to either 12 or 15 mm Hg depending on randomization. Both the patient and surgeon were blinded to the insufflation pressure. In post anesthesia care unit , patient reported pain scores were documented by nursing staff. Median immediate postoperative pain score and total required morphine milligram equivalents (MME) were recorded. On postop day one, participants were be asked to rate their pain with a numeric rating scale by a registered nurse. At 2 weeks postoperatively, participants were asked to rate their pain with a numeric rating scale and completed the Patient Global Impression of Improvement. At both visits, the clinical team member asked the patient how many narcotic tablets they have left to calculate total MME use outpatient. The clinical team member conducting these visits was blinded to randomization groups. Pain scores and patient responses were collected as well as demographics, clinical characteristics, surgery details, intraoperative outcomes, and 2 week postoperative outcomes. The investigators estimate the median numeric rating scale score in the immediate postoperative period to be 75 mm in the standard insufflation pressure group based on prior literature. The investigators calculated that 32 patients in each group are needed to detect a significant improvement of median numeric rating scale score to 60 mm in the experimental group. The investigators planned to enroll at least 64 participants to have 80% power to detect a 15 mm difference in scores between the two groups assuming a two-sided significance level of 5%. Assuming a 10% drop out rate, a total sample of 70 participants was recruited.

ELIGIBILITY:
Inclusion Criteria:

* Adult women scheduled for single port robotic sacrocolpopexy for uterovaginal or vaginal vault prolapse

Exclusion Criteria:

* Non-english speaking
* Inability to complete study questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Post anesthesia Care Unit Pain | 0 mins-4 hours after surgery
  Immediate after surgery in the post anesthesia care unit (PACU), patients were asked to rate their pain using a 100 point numeric rating scale (0 [no pain] to 100 [worst imaginable pain]). The PACU nurse routine asked pain score with routine vitals. The median score was recorded.

SECONDARY OUTCOMES:
Post anesthesia care unit morphine milligram equivalents | 0 mins-4 hours
  The total amount of morphine milligram equivalents the patient received in PACU was recorded.
Postoperative day one pain | 24 hours after surgery
  On postoperative day one telephone call, patients were asked to rate their pain using a 100 point numeric rating scale (0 [no pain] to 100 [worst imaginable pain]) by the clinical team member.
Postoperative day one morphine milligram equivalents | 24 hours after surgery
  On postoperative day one telephone call, patients were asked how many tablets of narcotics they had taken since discharge. Morphine milligram equivalents was then recorded.
Postoperative day 14 pain | 14 days after surgery
  At postoperative day 14 telemedicine visit, patients were asked to rate their pain using a 100 point numeric rating scale (0 [no pain] to 100 [worst imaginable pain]) by the clinical team member.
Postoperative day 14 morphine milligram equivalents | 14 days after surgery
  At postoperative day 14 telemedicine visit, patients were asked how many tablets of narcotics they had taken since discharge. Morphine milligram equivalents was then recorded.
Patient Global Impression of Improvement | 14 days after surgery
  At postoperative day 14 telemedicine visit, the patients were asked to complete the Patient Global Impression of Improvement (1 [very much improved] to 7 [very much worse]). Answers were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret G Mueller, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No